CLINICAL TRIAL: NCT00209001
Title: Efficacy of Acupuncture for Hot Flashes in Women Treated With Hormonal Therapy for Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator Peter Johnstone, MD relocated to another institution
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Keerthi Gogineni, Assistant Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0533-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham acupuncture therapy (Sham Comparator): Sham acupuncture therapy
  Interventions: Procedure: Sham acupuncture therapy
- Acupuncture (Active Comparator): Acupuncture
  Interventions: Procedure: Acupuncture
- Observation (No Intervention): Observation

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture using enhanced Ming Men technique for 20 minutes, twice during 1st week, then once during week 2, 3,and 4.
  Arms: Acupuncture
Procedure: Sham acupuncture therapy — Sham procedure will be insertion of 5 needles for 20 minutes provided twice during first week, then once per week thereafter.
  Arms: Sham acupuncture therapy

SUMMARY:
The purpose of this study is to determine if acupuncture is effective in relieving hot flashes in women treated with hormonal therapy for breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine if acupuncture is effective in relieving hot flashes in women treated with hormonal therapy for breast cancer.

Hormonal therapy is one of the most common treatments for breast cancer in women. Unfortunately, many women on hormonal therapy suffer from hot flashes (the sudden sensation of heat throughout the face, neck and chest, with or without shivering and sweating). Many medicines have been used to treat hot flashes, but no single medication has been found to work reliably.

Acupuncture has been shown to be effective for many conditions in Western medicine specifically for dry mouth in people who have received radiation to their head and neck, as well as for hot flashes in women during menopause (the "change of life"). In this study, we are investigating whether acupuncture is effective for women suffering hot flashes that result from their treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* History of breast cancer who have received hormonal therapy
* Personal history of hot flashes
* Patients will be accepted if receiving therapy with traditional allopathic medicines if their hot flashes have persisted after two months

Exclusion Criteria:

* Receiving therapy with traditional allopathic medicines for hot flashes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Define efficacy of acupuncture to points of the enhanced Ming Men technique for relief of hot flashes after hormonal therapy for breast cancer. | weekly evaluation up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johnstone, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States